CLINICAL TRIAL: NCT00203281
Title: Pharmacokinetic Evaluation of Plasmapheresis in Cross Match Positive or ABO Incompatible Kidney Allograft Recipients
Brief Title: Study to Evaluate the Amount of Medications That May be Removed From the Body During Plasmapheresis
Status: Withdrawn | Type: Observational
Why Stopped: funding withdrawn
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Other Study IDs: 03U.86
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2016-10-21 (Estimated); Status verified 2016-10

CONDITIONS: Kidney Transplantation; Plasmapheresis
Keywords: renal transplantation
MeSH Terms: interventions — Tacrolimus; Mycophenolic Acid; Daclizumab; Immunoglobulins, Intravenous; Plasmapheresis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: tacrolimus
Drug: mycophenolate mofetil
Drug: daclizumab
Drug: intravenous immune globulin
Procedure: plasmapheresis

SUMMARY:
Based on the limited amount of experience with plasmapheresis and CytoGam concomitant use, the researchers seek to evaluate the pharmacokinetics (drug absorption, distribution, and elimination) of this therapy. The researchers are also interested in evaluating the pharmacokinetics of the various immunosuppressant medications that patients will receive such as tacrolimus, mycophenolate mofetil and daclizumab.

DETAILED DESCRIPTION:
Kidney transplantation has emerged as a desired treatment of choice for patients with end stage renal disease. Although transplantation has become increasingly successful, there continues to be risks associated with it. Prior to performing a kidney transplant patients are cross-matched (a test to determine whether or not they have preformed antibodies to the donor). Preformed antibodies result from a previous pregnancy, blood or platelet transfusion or prior transplant. Performing a transplant in patients who have preformed antibodies against the donor generally results in hyperacute rejection (when the immune system attacks the new kidney). This hyperacute rejection usually results in kidney loss in a very high percentage of patients. Due to these consequences, pre-transplant cross-matching has emerged as a standard of care. Although hyperacute kidney loss has now been avoided, a large population of highly sensitized patients that has little hope of receiving a transplant has been identified.

A number of groups have studied methods to lower specific antibody levels in a variety of clinical settings. The two primary methods used today in transplantation are plasmapheresis (the separation of plasma from cells, and the removal of solutes, immune globulins, and medications) and administration of immune globulin therapy. Employing either of these techniques individually or jointly has substantially reduced acute rejection and improved kidney survival in these highly sensitized patients. The immune globulin treatments that have been studied have included large variations in dosage as well as differences in immune globulin products. The results from these small studies have not identified one therapy, product or dosage that could be considered standard of care.

The kidney transplant work-up also consists of matching ABO blood group between donor and recipient. Transplantation against the recipient blood group has resulted in very poor outcomes due to antibody mediated rejection (when the immune system attacks the kidney). However, due to the shortage of organs available for transplantation, the increasing number of patients awaiting a transplant and the favorable outcomes with live donor transplant, some transplant programs have developed protocols for transplanting against the recipient ABO blood group. These protocols are centered around plasmapheresis and treatment with immune globulin. As with the positive cross-match patients stated earlier, the standard of care has yet to be identified.

Dr. Lloyd Ratner, currently at Columbia University and former Chief of Transplant at Thomas Jefferson University Hospital and his former colleagues at Johns Hopkins University have studied the use of plasmapheresis in combination with Cytomegalovirus Immune Globulin Intravenous (CytoGam) to reverse a positive cross match and to transplant organs against ABO incompatible blood groups. This has enabled over 20 kidney transplants to be performed with patient and graft survival at one year being very similar to our traditional cross match negative and ABO compatible patients. These results are generally considered outstanding given the fact that antibody mediated rejection historically had a 75 to 100% incidence of graft loss.

The treatment protocol that is used consists of plasmapheresis treatments alternating with CytoGam infusions every other day for 3 to 9 treatments prior to transplantation and another 1-5 treatments after transplant. Plasmapheresis is increasingly performed to treat various infectious, immunological, metabolic and inherited diseases. In this procedure, plasma and cellular components of blood are separated and solutes in plasma, including drugs may be removed. Generally, a volume of 1 to 1.5 times the plasma volume is removed and replaced with an equivalent volume of crystalloid or colloid. The procedure removes solutes or drugs from the blood compartment and the tissue stores remain unaffected except for re-equilibration with decreasing plasma concentrations. After each plasmapheresis treatment patients receive an infusion of CytoGam which is used to "inactivate" the remaining antibody. However, it is not known to what extent subsequent treatments of plasmapheresis remove CytoGam that patients received only hours or days prior.

During the treatment phase with plasmapheresis patients also receive a number of other medications such as immunosuppressants for the prevention and treatment of graft rejection, antibiotics for prevention and treatment of infection and various other medications for related illnesses. The effects that plasmapheresis may have on removal of these medications is not known for many of these agents. This information would be helpful for the potential need to re-dose or give supplemental doses of medications. This is extremely important for the immunosuppressant medications since under-dosing of these agents may result in serious negative outcomes. Due to these many unknown aspects it would be useful to know the extent of drug removal during plasmapheresis treatments. This would enable more precise dosing and ultimately better patient care.

ELIGIBILITY:
Inclusion Criteria:

* Patient is a male or female.
* Age of 18-75.
* Patient must have the ability to provide informed consent.
* Positive cross-match with intended donor and/or ABO incompatible with intended donor.

Exclusion Criteria:

* Patients under the age of 18 or over the age of 75.
* Women that are currently pregnant.
* Patient has a history of any illness that, in the opinion of the investigator(s), might confound the results of the study or pose additional risk to the patient.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospital setting
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2003-02; Primary Completion 2009-09 (Estimated); Study Completion 2009-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Chaballa, PharmD, Principal Investigator — Thomas Jefferson University
Locations (2):
- United States (2):
  - Columbia University, New York, New York
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania